CLINICAL TRIAL: NCT04004221
Title: A Single-Arm, Multicenter Phase 2 Study of BGB-A317 in Patients With Previously Treated PD-L1+ Locally Advanced or Metastatic Urothelial Bladder Cancer
Brief Title: Study of Tislelizumab in Participants With Locally Advanced or Metastatic Urothelial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-204; CTR20170071 (Registry Identifier: Center for drug evaluation, CDE)
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced or Metastatic Urothelial Bladder Cancer
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab (Experimental): 200mg intravenously (IV) every 3 weeks(Q3W)
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — 200mg intravenously (IV) every 3 weeks (Q3W)
  Other Names: BGB-A317

SUMMARY:
This was a single-arm, multicenter, Phase 2 study to evaluate the efficacy and safety of the anti- programmed cell death-1(PD-1) monoclonal antibody BGB-A317 in participants with PD-L1+, locally advanced or metastatic Urothelial Bladder Cancer (UBC) who have progressed during or following a platinum-containing regimen

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with histologically or cytologically documented locally advanced or metastatic transitional cell carcinoma (TCC) of the urothelium
2. Disease progression during or following treatment with at least one platinum-containing regimen for inoperable locally advanced or metastatic urothelial carcinoma or disease recurrence
3. Participants must submit archival tumor tissue for determination of program death ligand-1 (PD-L1) expression and other biomarker analyses. PD-L1 expression will be assessed centrally, and participants who are tested as PD-L1 high are eligible.
4. Participants must have at least one measurable lesion as defined per RECIST version 1.1 assessed by the investigator
5. Male or female, aged ≥18 years on day of signing informed consent
6. Participants have voluntarily agreed to participate by giving written informed consent
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
8. Life expectancy ≥12 weeks
9. Participant must have adequate organ function as indicated by the following screening laboratory values obtained within 7 days prior to the first study treatment

   1. Absolute neutrophil count (ANC) ≥1.5×109/L
   2. Platelets ≥100×109/L
   3. Hemoglobin ≥9 g/dL or ≥5.6 mmol /L (Note: Criteria must be met without a transfusion within 14 days of obtaining the sample)
   4. Calculated creatinine clearance ≥ 30 milliliter (mL)/min (Cockcroft-Gault formula, see Appendix 5)
   5. Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN) (total bilirubin must be <4 X ULN for participants with Gilbert's syndrome)
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 X ULN OR ≤ 5 X ULN for participants with liver metastases
10. Female participants are eligible to enter and participate in the study if they are of:

    1. Non-childbearing potential (ie, physiologically incapable of becoming pregnant), including any female who i) Has had a hysterectomy ii) Has had a bilateral oophorectomy (ovariectomy) iii) Has had a bilateral tubal ligation iv) Is post menopausal (total cessation of menses for ≥1 year)
    2. Childbearing potential, has a negative serum pregnancy test at screening (within 7 days before the first investigational product administration), not be breast feeding, and agree to remain abstinent (refrain from heterosexual intercourse) or uses adequate contraceptive methods that result in a failure rate of <1% per year before study entry and throughout the study until 120 days after the last investigational product administration
11. Male participants are eligible to participate in the study if they are vasectomized or agree to use contraception during the study treatment period and for at least 120 days after the last dose of study drug

Key Exclusion Criteria:

1. History of severe hypersensitivity reactions to other humanized monoclonal antibodies
2. Prior active malignancy within 2 years prior to Cycle 1 Day 1.
3. Prior therapies targeting PD-1 or PD-L1.
4. Active brain or leptomeningeal metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments.
5. Participants with active autoimmune diseases or history of autoimmune diseases that may relapse should be excluded.
6. Participants should be excluded if they have conditions requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
7. Has history of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies
8. With severe chronic or active infections (including tuberculosis infection, etc) requiring systemic antibacterial, antifungal or antiviral therapy within 14 days prior to first dose of study drug.
9. With uncontrollable pleural effusion, pericardial effusion or ascites requiring pleurocentesis or abdominal tapping less than 4 weeks
10. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina
11. Known history of Human Immunodeficiency Virus (HIV)
12. Participants with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carrier with HBV deoxyribonucleic acid (DNA) ≥500 IU/mL (or 2.5 × 103 cps/mL), or active hepatitis C should be excluded. Participant with inactive hepatitis B surface antigen (HBsAg) carrier, active HBV infection with sustained anti-HBV suppression (HBV DNA <500 IU/mL or 2.5 × 103 cps/mL) and participants whose hepatitis C has been cured (hepatitis C virus [HCV] ribonucleic acid [RNA] is lower than detection limit) can be enrolled
13. Underlying medical conditions that, in the investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events (AEs)
14. Prior chemotherapy, radiotherapy, immunotherapy or any investigational therapies (including Chinese herbal medicine and Chinese patent medicines) used to control cancer within 2 weeks of Cycle 1 Day 1. AEs associated with these therapies must be Grade 0-1, baseline or stabilized (except for alopecia)
15. Prior allogeneic stem cell or solid organ transplant
16. Administration of a live or attenuated vaccine within 4 weeks prior to study drug administration
17. Major surgical procedure other than for diagnosis within 28 days prior to study drug administration

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (27):
- China (24):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Cancer Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Provincial Wenzhou Hospital of Zhejiang, Wenzhou, Zhejiang
- South Korea (3):
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
Upon request, and subject to certain criteria, conditions, and exceptions, BeiGene will provide access to individual de-identified participant data from BeiGene-sponsored global interventional clinical studies conducted for medicines for indications that have been approved or in programmes that have been terminated. BeiGene will also consider requests for the protocol, data dictionary, and statistical analysis plan. Data requests can be submitted to medicalinformation@beigene.com.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Ye D, Liu J, Zhou A, Zou Q, Li H, Fu C, Hu H, Huang J, Zhu S, Jin J, Ma L, Guo J, Xiao J, Park SH, Zhang D, Qiu X, Bao Y, Zhang L, Shen W, Bi F. Tislelizumab in Asian patients with previously treated locally advanced or metastatic urothelial carcinoma. Cancer Sci. 2021 Jan;112(1):305-313. doi: 10.1111/cas.14681. Epub 2020 Nov 6. PMID 33047430
- [Derived] Ye D, Desai J, Shi J, Liu SM, Shen W, Liu T, Shi Y, Wang D, Liang L, Yang S, Ma X, Jin W, Zhang P, Huang R, Shen Z, Zhang Y, Wu YL. Co-enrichment of CD8-positive T cells and macrophages is associated with clinical benefit of tislelizumab in solid tumors. Biomark Res. 2023 Mar 7;11(1):25. doi: 10.1186/s40364-023-00465-w. PMID 36879284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 113 participants were enrolled in 27 centers in China and 3 centers in South Korea. All efficacy evaluations were done until 16 September 2019, the primary data cut-off date. Safety evaluations were done until 11 March 2021, the study completion date.
Groups:
- Tislelizumab: Participants received 200mg tislelizumab intravenously (IV) every 3 weeks (Q3W) until disease progression or death
Period: Overall Study
Arm/Group | Tislelizumab
Started | 113
Completed | 0
Not Completed | 113
Not completed — Death | 89
Not completed — Withdrawal by Subject | 5
Not completed — Participants transferred to Long-Term Extension (LTE) study | 9
Not completed — Sponsor Decision | 9
Not completed — Participant refused to enter LTE | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set includes all participants who received any dose of Tislelizumab
Arm/Group | Tislelizumab
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 84
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 5
  China | 108

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by Independent Review Committee (IRC)
Description: ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) assessed by Independent Review Committee (IRC) using RECIST version 1.1
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: The Efficacy Evaluable Analysis Set includes all participants who received any dose of tislelizumab and had measurable disease per IRC according to RECIST version 1.1 at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tislelizumab: Participants received 200mg tislelizumab IV Q3W until disease progression or death
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Percentage of participants | 24.0 [16.20 to 33.41]
Statistical Analysis 1: Comparison: Tislelizumab; Test type: Other; p < 0.0001, Exact Binomial Test; 1-sided p-value was based on binomial exact test of Tislelizumab versus historical rate of 0.1

2. Secondary Outcome: Duration of Response (DOR) as Assessed by IRC
Description: DOR - defined as the time from the first determination of a confirmed objective response by IRC according to RECIST version 1.1 until the first documentation of progression or death, whichever comes first
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Efficacy Evaluable Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Months | NA [8.41 to NA] — NA = Not Estimable due to insufficient number of events

3. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by IRC
Description: PFS is defined as the time from the date of first dose of study drug to the date of first documentation of disease progression assessed by IRC using RECIST version 1.1 or death, whichever occurs first
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Efficacy Evaluable Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Months | 2.1 [2.04 to 3.15]

4. Secondary Outcome: Disease Control Rate (DCR) as Assessed by IRC
Description: DCR is defined as the percentage of participants who achieve CR, PR and stable disease (SD) assessed by IRC using RECIST version 1.1
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Efficacy Evaluable Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Percentage of participants | 38.5 [29.09 to 48.51]

5. Secondary Outcome: Overall Survival (OS)
Description: OS - defined as the time from the date of first dose of study drug until the date of death from any cause
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 113
Months | 9.8 [7.46 to 12.48]

6. Secondary Outcome: ORR as Assessed by the Investigators
Description: ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as assessed by the investigators per RECIST version 1.1 and immune related RECIST (irRECIST)
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Efficacy Evaluable Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Percentage of participants
  RECIST | 24.0 [16.20 to 33.41]
  irRECIST | 24.0 [16.20 to 33.41]

7. Secondary Outcome: DOR as Assessed by Investigators Per RECIST Version 1.1 and irRECIST
Description: DOR is defined as the time from the first determination of a confirmed objective response by the investigator according to RECIST version 1.1 and irRECIST until the first documentation of progression or death, whichever comes first
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Efficacy Evaluable Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Months
  RECIST | NA [8.31 to NA] — NA = Not Estimable due to insufficient number of events
  irRECIST | NA [8.31 to NA] — NA = Not Estimable due to insufficient number of events

8. Secondary Outcome: PFS as Assessed by Investigators Per RECIST Version 1.1 and irRECIST
Description: PFS is defined as the time from the date of first dose of study drug to the date of first documentation of disease progression assessed by the investigator according to RECIST version 1.1 and irRECIST until the first documentation of progression or death, whichever comes first
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Efficacy Evaluable Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Months
  RECIST | 2.1 [2.07 to 3.58]
  irRECIST | 2.6 [2.07 to 4.07]

9. Secondary Outcome: DCR as Assessed by Investigators Per RECIST Version 1.1 and irRECIST
Description: DCR is defined as the percentage of participants who achieve CR, PR and stable disease (SD) assessed by investigators per RECIST version 1.1 and irRECIST
Time Frame: From the date of first dose up to approximately 2 years and 2 months
Population: Efficacy Evaluable Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 104
Percentage of participants
  RECIST | 41.3 [31.77 to 51.42]
  irRECIST | 46.2 [36.33 to 56.20]

10. Secondary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE is defined as an adverse event (AE) that had an onset date or a worsening in severity from baseline pre-treatment) on or after the first dose of study drug up to 30 days following study drug .discontinuation. An SAE is any untoward medical occurrence that, at any dose that results in death or is life-threatening.
Time Frame: From the date of first dose until End of Study (approximately 3 years and 9 months)
Population: Safety Analysis Set
Measure: Number; unit: Number of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 113
Number of participants
  Participants with At Least 1 TEAE | 112
  Grade 3 or Higher | 64
  Serious TEAEs | 49

ADVERSE EVENTS:
Time Frame: From the date of first dose until end of study (approximately 3 years and 9 months)
Groups:
- Tislelizumab: Participants received 200mg tislelizumab intravenously Q3W until disease progression or death.
Arm/Group | Tislelizumab
All-Cause Mortality (participants affected / at risk) | 89/113
Serious Adverse Events (participants affected / at risk) | 49/113
Other Adverse Events (participants affected / at risk) | 110/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=113)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 3 (3)
Liver injury (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Optic nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Device occlusion (Product Issues) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=113)
Anaemia (Blood and lymphatic system disorders) | 44 (58)
Hyperthyroidism (Endocrine disorders) | 6 (7)
Hypothyroidism (Endocrine disorders) | 11 (19)
Abdominal distension (Gastrointestinal disorders) | 12 (15)
Abdominal pain (Gastrointestinal disorders) | 9 (9)
Constipation (Gastrointestinal disorders) | 25 (28)
Diarrhoea (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 13 (16)
Vomiting (Gastrointestinal disorders) | 10 (11)
Asthenia (General disorders) | 9 (12)
Fatigue (General disorders) | 10 (10)
Oedema peripheral (General disorders) | 8 (8)
Pyrexia (General disorders) | 22 (27)
Nasopharyngitis (Infections and infestations) | 10 (14)
Upper respiratory tract infection (Infections and infestations) | 11 (12)
Urinary tract infection (Infections and infestations) | 23 (33)
Alanine aminotransferase increased (Investigations) | 19 (25)
Aspartate aminotransferase increased (Investigations) | 22 (28)
Blood alkaline phosphatase increased (Investigations) | 15 (19)
Blood bilirubin increased (Investigations) | 8 (13)
Blood creatine phosphokinase MB increased (Investigations) | 7 (10)
Blood creatinine increased (Investigations) | 19 (21)
Blood lactate dehydrogenase increased (Investigations) | 10 (11)
Blood urea increased (Investigations) | 9 (12)
Gamma-glutamyltransferase increased (Investigations) | 8 (8)
Neutrophil count decreased (Investigations) | 6 (18)
Platelet count decreased (Investigations) | 6 (7)
Weight decreased (Investigations) | 7 (7)
White blood cell count decreased (Investigations) | 8 (15)
Decreased appetite (Metabolism and nutrition disorders) | 23 (27)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (9)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 (16)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 (24)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 21 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (16)
Dizziness (Nervous system disorders) | 6 (7)
Insomnia (Psychiatric disorders) | 6 (7)
Haematuria (Renal and urinary disorders) | 8 (9)
Proteinuria (Renal and urinary disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (34)
Rash (Skin and subcutaneous tissue disorders) | 17 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04004221/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT04004221/SAP_001.pdf